CLINICAL TRIAL: NCT01431768
Title: Clinical Validation of the Respirio Flu Test for the Rapid Identification of Influenza A/B in the Primary Health Setting
Brief Title: Validation of the Respirio Flu Test for the Rapid Identification of Influenza A/B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Respirio Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RESP11001
Record Dates: First submitted 2011-09-07; First posted 2011-09-12 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Influenza
Keywords: Influenza; Human; Orthomyxoviridae infections; RNA Virus Infections; Virus Diseases; Respiratory Tract infections; Respiratory Tract Diseases
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections; RNA Virus Infections; Virus Diseases; Respiratory Tract Infections; Respiratory Tract Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Respirio Flu Test — The Respirio Flu Test (RFT) is a rapid test for identifying whether a patient is infected with the Influenza A or B virus. The test separates the Influenza virus from the patient's nose blow sample and utilizes the same underlying technology as a pregnancy test (lateral flow/immuno-chromatography) to deliver a positive or negative result in less than 10 minutes. The RFT is easy to use, designed with a 3 step process similar to that of the home pregnancy test. Results are presented to the patient as a combination of different coloured lines, depending on whether the patient has Influenza A or B.

SUMMARY:
This is a open label, prospective, pair comparison, randomised, multi-centre trial. The primary aim of this study to is to clinically validate the sensitivity and specificity of the Respirio Flu Test (RFT) in detecting Influenza A as compared with (a) the best available rapid Influenza A test in the market Quidel QuickVue (QQV) and (b) the gold standard for identifying Influenza A infection Polymerase Chain Reaction (PCR).

The secondary aim is to clinically validate the sensitivity and specificity of the Respirio Flu Test (RFT) in detecting Influenza B as compared to QQV and PCR.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged between 7 and 80 years (inclusive);
2. Fever > 37.5 or a self-reported history of fever or feeling feverish (includes fever controlled by medication) in the absence of documented fever;
3. Cough or sore throat;
4. Rhinorrhea or nasal congestion;
5. ≤ 5 days from onset of clinical Influenza - Like Illness (ILI) symptoms;
6. Subject (or parent/guardian) capable and willing to give informed consent;
7. Subject provides written assent according to his/her age, if applicable.

Exclusion Criteria:

1. Recent craniofacial abnormality or injury (last 3 months);
2. Nasal or sinus surgery, including surgery to correct deviation of the nasal septum, within the previous 6 months;
3. Craniofacial abnormality, such as severe deviation of the nasal septum;
4. Onset of clinical Influenza - Like Illness (ILI) symptoms > 5 days;
5. Know history of allergic reaction to plastics or adhesives;
6. Subject (or parent/guardian) unwilling or unable to give informed consent.

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of Influenza A | Day 1

SECONDARY OUTCOMES:
Sensitivity and specificity of Influenza B | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Julie Todhunter, MBBS, Principal Investigator — Unaffliated
Locations (2):
- Australia (2):
  - Taringa 7 Day Medical Practice, Brisbane, Queensland
  - Capalaba Medical Centre, Brisbane, Queensland